CLINICAL TRIAL: NCT01731353
Title: FungiScope - A Global Emerging Fungal Infection Registry
Acronym: FungiScope
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Pfizer (Industry); Basilea Pharmaceutica (Industry); Cidara Therapeutics Inc. (Industry); F2G Biotech GmbH (Industry); Matinas Biopharma, Inc (Industry)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Dr. med., University of Cologne
Other Study IDs: Fungi001
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Invasive Fungal Disease
Keywords: invasive fungal infection; Web-based registry
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * fixed tissue
  * fungal culture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Emerging fungal infections: Web-based registry of invasive infections by emerging fungi

SUMMARY:
The objective of this registry is to broaden the knowledge on epidemiology, diagnostic procedures and clinical course of emerging invasive fungal infections.

DETAILED DESCRIPTION:
The specific objectives are:

1. To determine the fungal species causing invasive fungal infection in different parts of the world.
2. To determine the clinical pattern of disease and document procedures performed for confirmation of the diagnosis.
3. To describe the therapeutic regimens used and their efficacy.
4. To share clinical isolates among the contributors of Fungiscope.
5. To develop molecular biology tools for identification of strains in histopathologically proven invasive fungal infection.

ELIGIBILITY:
Inclusion Criteria:

* Cultural, histopathological, antigen or DNA evidence of invasive fungal infection

Exclusion Criteria:

* Infection due to Candida spp., Cryptococcus neoformans, Pneumocystis jiroveci
* Endemic fungal infection such as coccidioidomycosis or histoplasmosis
* Colonisation or other non-invasive infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Invasive infections caused by emerging fungi
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2003-03; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy of emerging fungal infections | At 90 days from diagnosis
  failure, stable disease, partial response or complete response

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A. Cornely, Professor, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Koehler P, von Stillfried S, Garcia Borrega J, Fuchs F, Salmanton-Garcia J, Pult F, Boll B, Eichenauer DA, Shimabukuro-Vornhagen A, Kurzai O, Boor P, Kochanek M, Cornely OA. Aspergillus tracheobronchitis in COVID-19 patients with acute respiratory distress syndrome: a cohort study. Eur Respir J. 2022 May 5;59(5):2103142. doi: 10.1183/13993003.03142-2021. Print 2022 May. PMID 35144992
- [Derived] Hassler A, Lieb A, Seidel D, Cesaro S, Greil J, Klimko N, Khostelidi S, Solopova G, Ogunc D, Duran Graeff L, Cornely OA, Vehreschild MJ, Lehrnbecher T. Disseminated Fusariosis in Immunocompromised Children-Analysis of Recent Cases Identified in the Global Fungiscope Registry. Pediatr Infect Dis J. 2017 Feb;36(2):230-231. doi: 10.1097/INF.0000000000001396. PMID 27846057
- [Derived] Marty FM, Ostrosky-Zeichner L, Cornely OA, Mullane KM, Perfect JR, Thompson GR 3rd, Alangaden GJ, Brown JM, Fredricks DN, Heinz WJ, Herbrecht R, Klimko N, Klyasova G, Maertens JA, Melinkeri SR, Oren I, Pappas PG, Racil Z, Rahav G, Santos R, Schwartz S, Vehreschild JJ, Young JH, Chetchotisakd P, Jaruratanasirikul S, Kanj SS, Engelhardt M, Kaufhold A, Ito M, Lee M, Sasse C, Maher RM, Zeiher B, Vehreschild MJGT; VITAL and FungiScope Mucormycosis Investigators. Isavuconazole treatment for mucormycosis: a single-arm open-label trial and case-control analysis. Lancet Infect Dis. 2016 Jul;16(7):828-837. doi: 10.1016/S1473-3099(16)00071-2. Epub 2016 Mar 9. PMID 26969258
- See also: FungiScope - A Global Emerging Fungal Infection Registry — http://www.fungiscope.net
- See also: FungiQuest - Search Engine for rare fungal infection — http://fungiquest.net/